CLINICAL TRIAL: NCT06046742
Title: A Phase I, Open-label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Effects of M1-c6v1 for Treatment of Patients with Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of Intravenous M1-c6v1 for Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-J01
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor
Keywords: M1-c6v1; Solid Tumor; Oncolytic Virus; VRT106

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- M1-c6v1 intravenous injection (Experimental): M1-c6v1 will be administered through IV drip
  Interventions: Biological: M1-c6v1

INTERVENTIONS:
Biological: M1-c6v1 — Intravenous drip administration

SUMMARY:
A Phase I Study of the Safety and Tolerability of M1-c6v1 Administered Via Intravenously for Treatment of Patients With Locally Advanced or Metastatic Solid Tumors

DETAILED DESCRIPTION:
This study is an open-label, dose-escalation clinical study which aims to evaluate the safety and tolerability of multiple IV injections of M1-c6v1 in subjects with locally advanced/metastatic solid tumors, as well as evaluating the biological distribution characteristics and biological effects of M1-c6v1 (i.e., virus tissue distribution and shedding characteristics), evaluating immunogenicity of M1-c6v1, and preliminarily exploring the anti-tumor effects of M1-c6v1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have diagnosis of locally advanced or metastatic solid tumors who are intolerable or refractory to the standard therapy.
2. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board -approved informed consent prior to performing any of the Screening Visit procedures.
3. Males and females at least 18 years of age, inclusive, at the Screening Visit.
4. Have at least one measurable lesion.
5. An Eastern Cooperative Oncology Group (ECOG) score of 0-1, 1 week before the first administration of IMP.
6. An estimated survival time of ≥ 12 weeks.

Exclusion Criteria:

1. Subject has a history of primary or acquired immunodeficient states, leukemia, lymphoma, acquired immunodeficiency syndrome (AIDS) or other clinical manifestations of infection with human immunodeficiency viruses, and those on immunosuppressive therapy.
2. Subject has received any anti-tumor treatment 4 weeks before using the IMP, including chemotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy.
3. Subject has received systemic glucocorticoids (prednisone >10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents within 14 days prior to first administration of IMP.
4. Subject has received immunomodulatory drugs, including but not limited to thymosin, IL-2, IFN, etc. within 14 days prior to first administration of IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of intravenous M1-c6v1 in Patients with advanced malignant tumors | About 2 years
  Monitor the incidence of adverse events (TEAEs) during the study.
Evaluate dose-limiting toxicities (DLTs) and determine the recommended phase 2 dose (RP2D) of single-agent intravenous administration of M1-c6v1. | About 2 years
  Incidence of DLT
Conduct a dose extension study to evaluate the safety and tolerability of intravenous administration of M1-c6v1 at maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) levels. | About 2 years
  Monitor the incidence of adverse events (TEAEs) during the study.

SECONDARY OUTCOMES:
Examine the biological distribution characteristics and shedding patterns of intravenously administered M1-c6v1. | About 2 years
  Measure the distribution and shedding of M1-c6v1 following intravenous injection by detecting its presence in blood, saliva, urine, nasal swabs, and feces using qPCR (quantitative polymerase chain reaction) method.
Assess the immunogenicity of intravenous administration of M1-c6v1. | About 2 years
  Detect the presence of neutralizing antibodies against M1-c6v1 and assess their titers, which represent the potency of the neutralizing antibodies, using the PD50 value.
Assess the anti-tumor effect of M1-c6v1, including objective response rate (ORR) and disease control rate (DCR) as efficacy indicators. | About 2 years
  Based on the specific tumor types, assess the ORR (Objective Response Rate) and DCR (Disease Control Rate) using RECIST (Response Evaluation Criteria in Solid Tumors) v1.1 or mRECIST (modified Response Evaluation Criteria in Solid Tumors) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhou Virotech Pharmaceutical Co., Ltd., Study Chair — Guangzhou Virotech Pharmaceutical Co., Ltd.
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: No